CLINICAL TRIAL: NCT07080216
Title: A Multicenter, Open-label, Dose-finding and Dose-expansion Phase I/II Study of ZG005 in Combination With Gecacitinib in Participants With Advanced Cervical Cancer
Brief Title: Study of ZG005 in Combination With Gecacitinib in Participants With Advanced Cervical Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Suzhou Zelgen Biopharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ZG005-JAK-003
Record Dates: First submitted 2025-07-14; First posted 2025-07-23 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-07

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PART 1（phaseⅠ） (Experimental): Part 1 is a dose exploratory study of ZG005 combined with gecaxitinib ± bevacizumab to evaluate the tolerability and safety of the combination regimen
  Interventions: Biological: ZG005; Drug: Gecacitinib; Biological: Bevacizumab
- PART 2（phase II） (Experimental): Part 2 is a dose expansion study to further evaluate the safety and preliminary efficacy of the combination regimen identified in Part 1
  Interventions: Biological: ZG005; Drug: Gecacitinib; Biological: Bevacizumab

INTERVENTIONS:
Biological: ZG005 — ZG005 20mg/kg, intravenous infusion(IV), once every 3 weeks (Q3W)
Drug: Gecacitinib — Part 1: Cohort A：Gecacitinib is administered continuously until the end of treatment; Cohort B：Gecacitinib is administered continuously from CnD1 to D14, and discontinued from CnD15 to D21；Part 2：Gecacitinib for dose exploratory stage will commence after the Recommended Phase 2 Dose (RP2D) is determined during the dose escalation stage.
Biological: Bevacizumab — Bevacizumab 7.5 mg/kg，intravenous infusion(IV), once every 3 weeks (Q3W)

SUMMARY:
This is a multicenter, open-label phase I/II study in patients with advanced cervical cancer designed to evaluate the safety, tolerability, and preliminary efficacy of ZG005 in combination with Gecacitinib ± bevacizumab.

ELIGIBILITY:
Inclusion Criteria:

* Fully understand the study and voluntarily sign the informed consent form.
* Female 18-75 years of age;
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
* Histologically or cytologically confirmed advanced cervical cancer, including squamous cell carcinoma, adenocarcinoma, or adenosquamous carcinoma.

Exclusion Criteria:

* Patients were deemed unsuitable for participating in the study by the investigator for any reasons.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-09-23 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Adverse Event (AE) | Up to 2 years
Objective response rate (ORR) | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jason Wu, Study Chair — Suzhou Zelgen Biopharmaceuticals Co.,Ltd
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China